CLINICAL TRIAL: NCT00691574
Title: Melatonin Levels in Sleep-disordered Smith-Magenis Syndrome: a Pilot Study
Brief Title: Melatonin Levels in Smith Magenis Syndrome (SMS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: eIRB 0668; n/a unfunded
Record Dates: First submitted 2008-05-30; First posted 2008-06-05 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Chromosome Disorders
Keywords: Smith-Magenis Syndrome; melatonin; circadian rhythm; sleep
MeSH Terms: conditions — Chromosome Disorders; Smith-Magenis Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Subjects will sit in front of a fluorescent bright light box while completing plasma samples to test for melatonin suppression in blood. This will be completed by both the SMS patient group and the control group of elderly individuals.
  Interventions: Device: Enviro-light artificial light box
- 1 (Experimental): Subjects will take up to 3 mg of melatonin daily and will complete frequent (every 2-4 weeks) of saliva and/or plasma sampling to test for a change in the timing of the body clock in response to the melatonin.
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — up to 3 mg, daily, for up to 1 year
  Arms: 1
Device: Enviro-light artificial light box — Subjects will sit in front of an artificial, fluorescent light box (10,000 lux) while completing 25-hours of hourly plasma samples. The light lux level will be well below that identified as safe by the FDA.
  Other Names: bright light treatment
  Arms: 2

SUMMARY:
The goal of this pilot project is to determine whether melatonin levels are disordered in patients with Smith-Magenis Syndrome (SMS) and whether melatonin treatment can correct abnormal circadian rhythms in SMS patients. In addition, the study investigates the effects of bright light in an elderly control population that exhibits low melatonin secretion.

DETAILED DESCRIPTION:
Participation involves 5 stages for SMS patients. First, Subjects will complete 4 sessions of 25-hour salivary or plasma sampling, with the last sampling occurring in front of a bright light box. Second, subjects will enroll in the melatonin treatment phase, involving a daily dose (up to 3 mg) for up to one year, with frequent (every 2-4 weeks) of 25-hour salivary or plasma sampling. During this stage, the subject and/or caregiver may also be asked to wear an activity wrist monitor, complete a daily sleep diary and behavioral questionnaires. Third, the subject may be asked to complete up to 3 25-hour sampling periods and take a melatonin pill on the same day to test how their body metabolizes the hormone, melatonin. The fourth stage is for subjects who are found to have an abnormal body rhythm. Subjects will complete a 25-hour plasma sampling period under bedrest to test for a hormone, Cortisol. The fifth stage is an optional 12-hour sleep analysis (polysomnography) to test for sleep disorders.

Control participants will complete an abbreviated protocol of the 3 baseline 25-hour sampling periods and 1 involving bright light exposure.

ELIGIBILITY:
Inclusion Criteria:

* Control participants:

  * 30 individuals: ages 55-85,
  * healthy without significant active medical problems.
* SMS patients:

  * 20 individuals: ages 3-50,
  * with a clinical diagnosis of Smith-Magenis Syndrome by a qualified Medical Geneticist, confirmed by cytogenetic analysis documenting deletion of chromosome band 17p11.2.

Exclusion Criteria:

* Control participants:

  * A current Axis I psychiatric or substance abuse disorder according to the DSM-IV Manual, abnormal heart, liver or kidney function, diagnoses of neurodegenerative or cerebrovascular disease (Alzheimer's disease, Parkinson's disease, stroke, etc.),
  * cognitive impairment (Mini-Mental State Score < 23) but without a formal diagnosis of dementia,
  * active symptoms of depression (Geriatric Depression Scale: 30 pt. version > 10),
  * current diagnosis of cataracts,
  * macular degeneration or retinopathy based on eye exam by an optometrist or ophthalmologist within the past year.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1998-09; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eilis Boudreau, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Sleep and Mood Disorders Lab, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] De Leersnyder H. Inverted rhythm of melatonin secretion in Smith-Magenis syndrome: from symptoms to treatment. Trends Endocrinol Metab. 2006 Sep;17(7):291-8. doi: 10.1016/j.tem.2006.07.007. Epub 2006 Aug 4. PMID 16890450
- [Background] Potocki L, Glaze D, Tan DX, Park SS, Kashork CD, Shaffer LG, Reiter RJ, Lupski JR. Circadian rhythm abnormalities of melatonin in Smith-Magenis syndrome. J Med Genet. 2000 Jun;37(6):428-33. doi: 10.1136/jmg.37.6.428. PMID 10851253

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Light Box: Subjects will sit in front of a fluorescent bright light box while completing plasma samples to test for melatonin suppression in blood. This will be completed by both the SMS patient group and the control group of elderly individuals.
  Enviro-light artificial light box: Subjects will sit in front of an artificial, fluorescent light box (10,000 lux) while completing 25-hours of hourly plasma samples. The light lux level will be well below that identified as safe by the FDA.
- Melatonin: Subjects will take up to 3 mg of melatonin daily and will complete frequent (every 2-4 weeks) of saliva and/or plasma sampling to test for a change in the timing of the body clock in response to the melatonin.
  Melatonin: up to 3 mg, daily, for up to 1 year
Period: Overall Study
Arm/Group | Light Box | Melatonin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Box | Melatonin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Circadian Phase Marker, as Measured by the Melatonin Levels in Serial Salivary and/or Plasma Samples
Time Frame: every 2-4 weeks throughout the entire study
Population: as for baseline characteristics
Arm/Group | Light Box | Melatonin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Polysomnography Sleep Disorder Assessment
Time Frame: 1 optional, 12-hour assessment towards the end of the study
Population: as for baseline characteristics
Arm/Group | Light Box | Melatonin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Wrist Actigraph Activity Levels as a Secondary Indicator of Circadian Phase
Time Frame: every 2-4 weeks throughout the entire study along with every Circadian Phase Marker assessment
Population: as for baseline characteristics
Arm/Group | Light Box | Melatonin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Light Box | Melatonin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analyses were not completed because, a unique provision in the American Recovery and Reinvestment Act (ARRA) of 2009 funding source unexpectedly prevented approval of a second year no-cost-extension in which completion of analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No